CLINICAL TRIAL: NCT04288791
Title: Evaluation of the Clinical Performance of Reinforced Glass Ionomer Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nessma Mohamed Mahmoud Sedky, Principle Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC16-033
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equia Forte Fil (Experimental)
  Interventions: Other: Equia Forte Fil; Other: Zirconomer Improved
- Zirconomer Improved (Experimental)
  Interventions: Other: Equia Forte Fil; Other: Zirconomer Improved

INTERVENTIONS:
Other: Equia Forte Fil — Glass hybrid innovation achieved through the introduction of ultrafine, highly reactive glass particles dispersed with conventional GI. The restoration is coated with Equia Forte coat which incorporates multi-functional monomer producing a tougher resin matrix. This system is designed as alternative of amalgam in posterior teeth.
Other: Zirconomer Improved — Zirconia reinforced GI, Glass Polyalkenoate restoration; it is designed to exhibit high strength where the glass component of this GI undergoes finely controlled micronization to achieve optimum particle size and characteristics .

SUMMARY:
This study is conducted to evaluate the clinical performance of class I reinforced glass ionomer restorations (Zirconomer Improved and Equia Forte Fil)

ELIGIBILITY:
Inclusion Criteria:

* Normal occlusal relation with normal dentition.
* Absence of pain from the tooth to be restored.
* Absence of any active periodontal and pulpal diseases from the tooth to be restored.
* Medium-sized (buccolingually and mesio-distally) occlusal carious lesions extending into dentin.

Exclusion Criteria:

* Patients with a history of tooth sensitivity.
* Patients with bruxism.
* Defective restorations adjacent or opposing to the tooth.
* Abutment teeth used for fixed or removable prosthesis.
* Patients who refused to sign the consent form.
* Inability to return to recall appointments

Ages: 20 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical Performance of the restoration | 6 months
  Success Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Faculty of Dentistry For Girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided